CLINICAL TRIAL: NCT01279850
Title: SPECIAL INVESTIGATION OF LONG TERM USE OF LYRICA(REGULATORY POST MARKETING COMMITMENT PLAN)
Brief Title: Safety And Efficacy In Long Term Use Of Lyrica (Regulatory Post Marketing Commitment Plan)
Acronym: RAINBOW-L
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081262
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Neuropathic Pain
Keywords: Lyrica; Regulatory Post Marketing Commitment Plan; Safety; Neuropathic Pain; Post Marketing Surveillance
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin; Capsules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregabalin (Lyrica) capsule: Patients administered "Pregabalin capsule".
  Interventions: Drug: Pregabalin (Lyrica) capsule

INTERVENTIONS:
Drug: Pregabalin (Lyrica) capsule — Lyrica® Capsules depending on the investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dosage for oral use begins at 150 mg/day of pregabalin in twice daily, and should be gradually increased to 300 mg/day over 1 week or more and should be orally administered twice daily. Dosage should be adjusted, depending on age or symptoms. However, the daily maximum dose should not be beyond 600 mg, and should be orally administered twice daily".
  Other Names: Lyrica® Capsules 25 mg, Lyrica® Capsules 75 mg, Lyrica® Capsules 150 mg

SUMMARY:
The objective of this investigation is to evaluate the safety and efficacy of long term use with Lyrica in medical practice. Also, occurrence of unknown and known adverse drug reactions (ADRs) in subjects treated with Lyrica will be monitored during the survey period, and whether an additional treatment outcome investigation and/or a post-marketing clinical study is required in the future will be determined.

DETAILED DESCRIPTION:
Patients who fulfill criteria below:

1. Patients who have previously enrolled in A0081261.
2. Patients who have been administered Lyrica for more than 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered by Lyrica for over 52 weeks in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Lyrica.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A0081262 prescribes the Lyrica capsule.
  And the patients who are administered Lyrica for over 52 weeks (MAX 104 weeks).
Sampling Method: Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081262&StudyName=Safety%20And%20Efficacy%20In%20Long%20Term%20Use%20Of%20Lyrica%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- LYRICA Capsules (Pregabalin): Participants who received LYRICA Capsules as indicated in the approved local product document were observed from the start of the treatment to Week 104 at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | LYRICA Capsules (Pregabalin)
Started | 891
Completed | 800 (Number of participants whose survey form were collected and included in analyses is shown.)
Not Completed | 91
Not completed — Protocol Violation | 50
Not completed — No Drug Administration Information | 7
Not completed — No Visit After Treatment | 34

BASELINE CHARACTERISTICS:
Population: Among 891 participants whose survey form was collected, a total of 91 participants were excluded from the baseline analysis population due to following reasons: protocol violation (50 participants), no drug administration information (7 participants), and no visit after treatment (34 participants).
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 267
  ≥65 years | 533
Sex/Gender, Customized [Number; unit: Participants]
  Male | 358
  Female | 442
Race/Ethnicity, Customized [Number; unit: Participants]
  Race and Ethnicity Not Collected | 800

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to Week 104 at maximum
Population: The analysis population for this outcome measure was the baseline analysis population, which comprised of participants who satisfied the criteria of safety analysis population and had received LYRICA Capsules at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Percentage of Participants | 12.75

2. Secondary Outcome: Percentage of Participants With Serious Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to Week 104 at maximum
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Percentage of Participants | 0.25

3. Secondary Outcome: Percentage of Participants With Adverse Drug Reaction Unexpected From Japanese Package Insert
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to Week 104 at maximum
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Percentage of Participants | 0.50

4. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Peripheral Edema or Other Edema-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to peripheral edema or other edema-related events was evaluated.
Time Frame: From Week 1 to Week 104 at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Participants | 14

5. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Dizziness, Somnolence, Loss of Consciousness, Syncope, and Potential for Accidental Injury
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to dizziness, somnolence, loss of consciousness, syncope, and potential for accidental injury was evaluated.
Time Frame: From Week 1 to Week 104 at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Participants | 65

6. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Vision-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to vision-related events was evaluated.
Time Frame: From Week 1 to Week 104 at maximum
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 800
Participants | 4

7. Secondary Outcome: Clinical Effectiveness Rate
Description: Clinical effectiveness of LYRICA Capsules was determined by the physician based on the following categories: (1) effective, (2) ineffective, or (3) impossible to judge at Week 104 of the treatment. Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of the analysis population, was presented along with the corresponding 2-sided 95% CI.
Time Frame: At Week 104
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of clinical effectiveness was available and who satisfied the inclusion criteria among the baseline analysis population. Of these, participants evaluated as "impossible to judge" were excluded from the analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 777
Percentage of Participants | 91.0 [88.8 to 93.0]

8. Secondary Outcome: Change From Baseline in Participant-rated Pain Score at Week 104
Description: The pain experienced at Week 104 during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (no pain) to 10 (the most severe pain possible). Mean change from baseline in participant-rated pain score at Week 104 was presented along with standard deviation.
Time Frame: Baseline and at Week 104
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of participant-rated pain score was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 113
Units on a scale | -4.4 (2.14)

9. Secondary Outcome: Change From Baseline in Participant-rated Sleep Interference Score at Week 104
Description: The sleep interference (inability to sleep because of pain) experienced at Week 104 during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (no disturbance) to 10 (totally unable to sleep because of pain). Mean change from baseline in participant-rated sleep interference score at Week 104 was presented along with standard deviation.
Time Frame: Baseline and at Week 104
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of participant-rated sleep interference score was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 104
Units on a scale | -3.9 (2.54)

10. Secondary Outcome: Patient's Impression (PGIC) at Week 104
Description: The patient's impression (patient global impression of change [PGIC]) at Week 104, as compared to the baseline condition (including the first day of treatment), was rated by participants on a 7-grade scale.
Time Frame: At Week 104
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of PGIC was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 791
Participants
  Markedly improved | 95
  Improved | 223
  Slightly improved | 183
  Unchanged | 71
  Slightly worsened | 3
  Worsened | 2
  Markedly worsened | 0
  Not assessed | 214

11. Secondary Outcome: Physician's Impression (CGIC) at Week 104
Description: The physician's impression (clinical global impression of change [CGIC]) at Week 104, as compared to the baseline condition (including the first day of treatment), was rated by the physician on a 7-grade scale.
Time Frame: At Week 104
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of CGIC was available and who satisfied the inclusion criteria among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 791
Participants
  Markedly improved | 108
  Improved | 275
  Slightly improved | 179
  Unchanged | 93
  Slightly worsened | 7
  Worsened | 0
  Markedly worsened | 0
  Not assessed | 129

ADVERSE EVENTS:
Time Frame: From Week 1 to Week 104 at maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | LYRICA Capsules (Pregabalin)
All-Cause Mortality (participants affected / at risk) | 7/800
Serious Adverse Events (participants affected / at risk) | 22/800
Other Adverse Events (participants affected / at risk) | 153/800
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=800)
Pneumonia (Infections and infestations) | 2
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Brain oedema (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Asthenia (General disorders) | 1
Condition aggravated (General disorders) | 1
Disease progression (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 1
Sudden death (General disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=800)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 4
Abnormal sensation in eye (Eye disorders) | 1
Cataract (Eye disorders) | 2
Conjunctivitis allergic (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Face oedema (General disorders) | 4
Oedema (General disorders) | 5
Oedema peripheral (General disorders) | 17
Peripheral swelling (General disorders) | 1
Thirst (General disorders) | 3
Alcoholic liver disease (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Pyoderma (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 5
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose fluctuation (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 8
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 38
Dysgeusia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 36
Syncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 6
Panic disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Fixed eruption (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Essential hypertension (Vascular disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Intermittent claudication (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-01-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT01279850/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT01279850/SAP_001.pdf